CLINICAL TRIAL: NCT02566759
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single and Multiple Doses of TAK-831 in Healthy Subjects
Brief Title: A TAK-831-1001, Single and Multiple Rising Dose Study in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by Takeda due to the discomfort observed in the study participants from the CSF collection procedure in Part 3 of the study.
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TAK-831-1001; 2015-002295-24 (EudraCT Number); U1111-1168-6568 (Registry Identifier: WHO); 15/SC/0412 (Registry Identifier: NRES)
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia, Cerebellar Ataxia
Keywords: Drug therapy
MeSH Terms: conditions — Schizophrenia; Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- Part 1, Cohort 1: TAK-831 100 mg (Experimental): TAK-831 100 milligram (mg), suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 1, Cohort 2: TAK-831 250 mg (Experimental): TAK-831 250 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 1, Cohort 3: TAK-831 500 mg (Experimental): TAK-831 500 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 1, Cohort 4: TAK-831 30 mg (Experimental): TAK-831 30 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 1, Cohort 5: TAK-831 750 mg (Experimental): TAK-831 750 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 1, Cohort 6: TAK-831 10 mg (Experimental): TAK-831 10 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 2, Cohort 1: TAK-831 30 mg (Experimental): TAK-831 30 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1 and once daily from Days 4 to 16.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 2, Cohort 2: TAK-831 100 mg (Experimental): TAK-831 100 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1 and once daily from Days 4 to 16.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 2, Cohort 3: TAK-831 200 mg (Experimental): TAK-831 200 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1 and once daily from Days 4 to 16.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 2, Cohort 4: TAK-831 400 mg (Experimental): TAK-831 400 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once on Day 1 and once daily from Days 4 to 16.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 3, Cohort 1: TAK-831 400 mg (Experimental): TAK-831 400 mg, suspension, orally or TAK-831 placebo-matching suspension, orally, once daily from Days 1 to 14.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Placebo
- Part 4:TAK-831(Tablet Fasted+ Tablet Fed + Suspension Fasted) (Experimental): TAK-831 100 mg, tablet, orally, once after an overnight fast of at least 10 hours on Day 1 of Period 1, followed by a washout interval of 5 days, further followed by TAK-831 100 mg, tablet, orally, once 30 minutes after starting a high fat meal on Day 1 of Period 2, followed by a washout interval of 5 days, further followed by TAK-831 100 mg, suspension, orally, once after an overnight fast of at least 10 hours on Day 1 of Period 3.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Tablet
- Part 4:TAK-831(Tablet Fed + Tablet Fasted + Suspension Fasted) (Experimental): TAK-831 100 mg, tablet, orally, once 30 minutes after starting a high fat meal on Day 1 of Period 1, followed by a washout interval of 5 days, further followed by TAK-831 100 mg, tablet, orally, once after an overnight fast of at least 10 hours on Day 1 of Period 2, followed by a washout interval of 5 days, further followed by TAK-831 100 mg, suspension, orally, once after an overnight fast of at least 10 hours on Day 1 of Period 3.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Tablet
- Part 4:TAK-831(Suspension Fasted+ Tablet Fed + Tablet Fasted) (Experimental): TAK-831 100 mg, suspension, orally, once after an overnight fast of at least 10 hours on Day 1 of Period 1, followed by a washout interval of 5 days, further followed by TAK-831 100 mg, tablet, orally, once 30 minutes after starting a high fat meal on Day 1 of Period 2, followed by a washout interval of 5 days, further followed by TAK-831 100 mg, tablet, orally, once after an overnight fast of at least 10 hours on Day 1 of Period 3.
  Interventions: Drug: TAK-831 Oral Suspension; Drug: TAK-831 Tablet

INTERVENTIONS:
Drug: TAK-831 Oral Suspension — TAK-831 oral suspension.
Drug: TAK-831 Placebo — TAK-831 placebo-matching oral suspension.
  Arms: Part 1, Cohort 1: TAK-831 100 mg; Part 1, Cohort 2: TAK-831 250 mg; Part 1, Cohort 3: TAK-831 500 mg; Part 1, Cohort 4: TAK-831 30 mg; Part 1, Cohort 5: TAK-831 750 mg; Part 1, Cohort 6: TAK-831 10 mg; Part 2, Cohort 1: TAK-831 30 mg; Part 2, Cohort 2: TAK-831 100 mg; Part 2, Cohort 3: TAK-831 200 mg; Part 2, Cohort 4: TAK-831 400 mg; Part 3, Cohort 1: TAK-831 400 mg
Drug: TAK-831 Tablet — TAK-831 tablet.
  Arms: Part 4:TAK-831(Suspension Fasted+ Tablet Fed + Tablet Fasted); Part 4:TAK-831(Tablet Fasted+ Tablet Fed + Suspension Fasted); Part 4:TAK-831(Tablet Fed + Tablet Fasted + Suspension Fasted)

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics (PK) of single and multiple rising doses of TAK-831 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831. TAK-831 is being tested to treat participant who have schizophrenia and cerebellar ataxia. This study will look at the PK, safety and tolerability of TAK-831 in healthy participants. The study will enroll approximately 120 participants. The study will include 4 parts: Part 1 (single-rising dose [SRD]), Part 2 (SRD/multiple-rising dose [MRD]), Part 3 (MRD) and Part 4 (relative bioavailability study). Participants will be randomly assigned (by chance, like flipping a coin) to receive either active drug TAK-831 or placebo which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Part 1, Cohort 1: single dose of TAK-831 100 mg
* Part 1, Cohort 2: single dose of TAK-831 250 mg
* Part 1, Cohort 3: single dose of TAK-831 500 mg
* Part 1, Cohort 4: single dose of TAK-831 30 mg
* Part 1, Cohort 5: single dose of TAK-831 750 mg
* Part 1, Cohort 6: single dose of TAK-831 10 mg
* Part 2, Cohort 1: single dose of TAK-831 30 mg
* Part 2, Cohort 2: single dose of TAK-831 100 mg
* Part 2, Cohort 3: single dose of TAK-831 200 mg
* Part 2, Cohort 4: single dose of TAK-831 400 mg
* Part 3, Cohort 1: TAK-831 400 mg
* Part 4: TAK-831 100 mg (Tablet Fasted + Tablet Fed + Suspension Fasted)
* Part 4: TAK-831 100 mg (Tablet Fed + Tablet Fasted + Suspension Fasted)
* Part 4: TAK-831 100 mg (Suspension Fasted+ Tablet Fed + Tablet Fasted)

Dosing with TAK-831 will progress into study Part 2, 3 and 4, only after review of all available safety, tolerability, and PK data collected in Cohorts 1 to 6 of the Study Part 1. This single center trial will be conducted in the United Kingdom. The overall time to participate in this study is approximately up to 58 days. Participants will be admitted in the clinic for the up to 20 days, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

The study was terminated by Takeda due to the discomfort observed in the study participants from the CSF collection procedure in Part 3 of the study, hence it is was not feasible to collect further CSF samples that were required to meet the exploratory objectives of the study. Part 1, 2 and 4 of the study were completed as planned.

ELIGIBILITY:
Inclusion Criteria:

1. Should be capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Healthy male or female aged between 18 to 55 years- Weighing at least 45 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2).
4. Male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
5. Female participant with no childbearing potential, defined as a participant that has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who is post menopausal (defined as continuous amenorrhea of at least 2 years and follicle-stimulating hormone [FSH] greater than [>] 40 international units per liter [IU/L]).

Exclusion Criteria:

1. Received any investigational compound within 3 months prior to randomization.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Has uncontrolled, clinically significant neurological (including seizure disorders), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality.
4. Has a known hypersensitivity to any component of the formulation of TAK-831.
5. Female participant is of childbearing potential.
6. Has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in.
7. History of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or 1 single measure of spirits or 1 small glass of wine.
8. Has taken any excluded medication, supplements, or food products during the time periods listed in the excluded medications and dietary products.
9. Female participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
10. Male participant intending to donate sperm during the course of this study or for 12 weeks after the last dose of study medication.
11. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma, hypoxemia, hypertension, seizures, or allergic skin rash.
12. Has a QT interval with Fridericia's correction method (QTcF) >450 millisecond (msec) (males) or >470 msec (females) or PR outside the range of 120 to 220 msec, confirmed with one repeat testing, at the screening visit or check-in (Day -2).
13. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention.
14. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
15. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody/antigen at Screening.
16. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in. Cotinine test is positive at Screening or Check-in.
17. Has poor peripheral venous access.
18. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to first dose of medication.
19. Has a Screening or Check-in abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator or designee.
20. Has a supine blood pressure outside the ranges of 90 to 140 millimeter of mercury (mm Hg) for systolic and 50 to 90 mm Hg for diastolic, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in.
21. Has a resting heart rate outside the range 40 to 100 bpm confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in.
22. Has abnormal Screening or check-in laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
23. Has a risk of suicide according to the Investigator's clinical judgment (example, per The Columbia Suicide Severity Rating Scale [C-SSRS]), or has scored "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior", if this behaviour occurred in the past 2 years.
24. Has received TAK-831 in a previous clinical study.
25. Participant is vegan or vegetarian (Part 4 only - food effect).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-09-23; Primary Completion 2016-06-09 (Actual); Study Completion 2016-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 23 September 2015 to 12 July 2016.
Pre-assignment Details: Healthy participants were enrolled in 4 part study to receive TAK-831: single rising dose (SRD) in Part 1; SRD/multiple rising dose (MRD) in Part 2; MRD in Part 3; relative bioavailability(rBA) in 3-sequence crossover in Part 4. Part 3 was terminated due to discomfort observed in participants from the cerebrospinal fluid (CSF) collection procedure.
Groups:
- Part 1: Placebo Pooled: TAK-831 placebo-matching suspension, orally, once on Day 1.
- Part 1: TAK-831 10 mg: TAK-831 10 milligram (mg), suspension, orally, once on Day 1.
- Part 1: TAK-831 30 mg: TAK-831 30 mg, suspension, orally, once on Day 1.
- Part 1: TAK-831 100 mg: TAK-831 100 mg, suspension, orally, once on Day 1.
- Part 1: TAK-831 250 mg: TAK-831 250 mg, suspension, orally, once on Day 1.
- Part 1: TAK-831 500 mg: TAK-831 500 mg, suspension, orally, once on Day 1.
- Part 1: TAK-831 750 mg: TAK-831 750 mg, suspension, orally, once on Day 1.
- Part 2: Placebo Pooled: TAK-831 placebo-matching suspension, orally, once on Day 1 and Days 4-16.
- Part 2: TAK-831 30 mg: TAK-831 30 mg, suspension, orally, once on Day 1 and Days 4-16.
- Part 2: TAK-831 100 mg: TAK-831 100 mg, suspension, orally, once on Day 1 and Days 4-16.
- Part 2: TAK-831 200 mg: TAK-831 200 mg, suspension, orally, once on Day 1 and Days 4-16.
- Part 2: TAK-831 400 mg: TAK-831 400 mg, suspension, orally, once on Day 1 and Days 4-16.
- Part 3: Placebo: TAK-831 placebo-matching suspension, orally, once daily on Days 1-14.
- Part 3: TAK-831 400 mg: TAK-831 400 mg, suspension, orally, once daily from Days 1-14.
- Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted): TAK-831 100 mg, tablet, orally, in fasted state, once on Day 1 of Period 1, followed by a 5-day washout period, further followed by TAK-831 100 mg, tablet, orally, in fed state, once on Day 1 of Period 2, followed by a 5-day washout period, further followed by TAK-831 100 mg, suspension, orally, in fasted state, once on Day 1 of Period 3.
- Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted): TAK-831 100 mg, tablet, orally, in fed state, once on Day 1 of Period 1, followed by a 5-day washout period, further followed by TAK-831 100 mg, tablet, orally, in fasted state, once on Day 1 of Period 2, followed by a 5-day washout period, further followed by TAK-831 100 mg, suspension, orally, in fasted state, once on Day 1 of Period 3.
- Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted): TAK-831 100 mg, suspension, orally, in fasted state, once on Day 1 of Period 1, followed by a 5-day washout period, further followed by TAK-831 100 mg, tablet, orally, in fed state, once on Day 1 of Period 2, followed by a 5-day washout interval, further followed by TAK-831 100 mg, tablet, orally, in fasted state, once on Day 1 of Period 3.
Period: All Parts
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted) | Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted) | Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted)
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 8 | 8 | 8
Completed | 12 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 5 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 8 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 6 (Participants from Part 1 and 2 did not continue in the washout period of Part 4 (crossover part).) | 0 | 0 | 8 (Only participants of Part 4 continued in next period.) | 8 (Only participants of Part 4 continued in next period.) | 8 (Only participants of Part 4 continued in next period.)
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Washout Crossover Period (Part 4:5 Days)
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted) | Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted) | Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Treatment (Part 4: 1 Day)
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted) | Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted) | Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout Crossover Period (Part 4:5 Days)
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted) | Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted) | Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Treatment (Part 4: 1 Day)
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted) | Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted) | Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 (Tablet Fasted+Tablet Fed+Suspension Fasted) | Part 4: TAK-831 (Tablet Fed+Tablet Fasted+Suspension Fasted) | Part 4: TAK-831 (Suspension Fasted+Tablet Fed+Tablet Fasted) | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 8 | 8 | 8 | 110
Age, Customized [Number; unit: participants]
  18 to 55 years | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 8 | 8 | 8 | 110
Sex/Gender, Customized [Number; unit: participants]
  Male | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 8 | 8 | 8 | 110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7
  White | 10 | 5 | 5 | 5 | 5 | 6 | 5 | 6 | 4 | 5 | 5 | 6 | 1 | 4 | 6 | 7 | 8 | 93
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 8 | 8 | 8 | 110
Smoking History [Number; unit: participants]
  Never smoked | 8 | 4 | 5 | 5 | 3 | 3 | 6 | 5 | 5 | 5 | 4 | 5 | 1 | 4 | 8 | 5 | 6 | 82
  Ex-smoker | 4 | 2 | 1 | 1 | 3 | 3 | 0 | 3 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 3 | 2 | 28
Alcohol history [Number; unit: participants]
  Never drunk | 3 | 1 | 3 | 2 | 1 | 1 | 4 | 3 | 4 | 3 | 0 | 0 | 1 | 3 | 2 | 1 | 1 | 33
  Current drinker | 9 | 5 | 3 | 4 | 5 | 5 | 2 | 5 | 2 | 3 | 6 | 6 | 0 | 2 | 6 | 7 | 7 | 77
Caffeine Consumption [Number; unit: participants]
  Caffeine consumption | 10 | 6 | 4 | 5 | 5 | 4 | 6 | 3 | 3 | 4 | 4 | 4 | 1 | 3 | 8 | 4 | 4 | 78
  No caffeine consumption | 2 | 0 | 2 | 1 | 1 | 2 | 0 | 5 | 3 | 2 | 2 | 2 | 0 | 2 | 0 | 4 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to 30 days after the last dose of study drug (Part 1 Day 31, Part 2 Day 46, Part 3 Day 44 and Part 4 Day 43)
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Part 4: TAK-831 100 mg Tablet Fasted: TAK-831 100 mg, tablet, orally, once in fasted state on Day 1 of either Period 1, 2 or 3.
- Part 4: TAK-831 100 mg Tablet Fed: TAK-831 100 mg, tablet, orally, once in fed state on Day 1 of either Period 1, 2 or 3.
- Part 4: TAK-831 100 mg Suspension Fasted: TAK-831 100 mg, suspension, orally, once in fasted state on Day 1 of either Period 1, 2 or 3.
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 23 | 23 | 24
percentage of participants | 50.0 | 33.3 | 33.3 | 33.3 | 16.7 | 50.0 | 66.7 | 75.0 | 83.3 | 100.0 | 33.3 | 83.3 | 100.0 | 100.0 | 21.7 | 13.0 | 16.7

2. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Description: Clinical laboratory tests included hematology, serum chemistry and urinalysis.
Time Frame: Baseline up to Day 15 in Part 1, Day 30 in Part 2, Day 28 in Part 3 and Day 25 in Part 4
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 23 | 23 | 24
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 33.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Description: Markedly abnormal criteria for vital signs measurement was assessed. The lower criteria and upper criteria for abnormality are as follow: systolic blood pressure at less than (<) 85 millimeter of mercury (mm Hg) to greater than (>) 180 mm Hg; diastolic blood pressure < 50 mm Hg to >110 mm Hg; pulse rate <50 bpm to >120 bpm; Temperature <35.6 degree Celsius to >37.7 degree Celsius.
Time Frame: Baseline up to Day 15 in Part 1, Day 30 in Part 2, Day 28 in Part 3 and Day 25 in Part 4
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 23 | 23 | 24
percentage of participants
  < lower criteria | 50.0 | 50.0 | 16.7 | 16.7 | 0 | 33.3 | 16.7 | 87.5 | 66.7 | 83.3 | 33.3 | 83.3 | 100.0 | 60.0 | 13.0 | 17.4 | 29.2
  > greater criteria | 8.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 33.3 | 0 | 20.0 | 4.3 | 8.7 | 12.5

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post Dose
Description: Markedly abnormal criteria for ECG was assessed. The lower cut-off point criteria and upper cut-off point criteria are as follow: heart rate <50 beats per minute (bpm) to >120 bpm; PR interval less than or equal to (<=) 80 millisecond (msec) to greater than or equal to (>=) 200 msec; QRS interval <=80 msec to >=180 msec; QT interval <=300 msec to >=460 msec; QTcB interval <=300 msec to >=500 msec or >=30 msec change from baseline and >=450 msec; QT interval with Fridericia's correction method (QTcF) interval <=50 msec to >=500 msec or >=30 msec change from baseline and >=450 msec.
Time Frame: Baseline up to Day 15 in Part 1, Day 30 in Part 2, Day 28 in Part 3 and Day 25 in Part 4
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 1 | 5 | 23 | 23 | 24
percentage of participants
  < lower cut-off point criteria | 41.7 | 33.3 | 16.7 | 50.0 | 16.7 | 33.3 | 16.7 | 37.5 | 33.3 | 50.0 | 0 | 16.7 | 0 | 20.0 | 13.0 | 21.7 | 16.7
  > upper cut-off point criteria | 8.3 | 50.0 | 0 | 16.7 | 0 | 33.3 | 16.7 | 25.0 | 50.0 | 16.7 | 16.7 | 16.7 | 0 | 0 | 8.7 | 13.0 | 12.5

5. Secondary Outcome: Part 1, 2 and 4: Cmax: Maximum Observed Plasma Concentration for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours in Part 1 and up to 72 hours in Part 2 and 4) post-dose
Population: The PK set included all participants with at least 1 estimable PK parameter for TAK-831.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 23 | 23 | 24
nanogram per milliliter (ng/mL) | 90.7 (26.95) | 313.3 (121.97) | 567.7 (218.76) | 905.8 (329.53) | 1304.5 (402.89) | 2121.7 (554.92) | 167.1 (39.95) | 467.2 (84.36) | 1087.3 (398.76) | 1095.5 (236.86) | 216.0 (104.68) | 377.7 (175.90) | 594.1 (288.77)
Statistical Analysis 1: Comparison: Part 1: TAK-831 10 mg vs Part 1: TAK-831 30 mg vs Part 1: TAK-831 100 mg vs Part 1: TAK-831 250 mg vs Part 1: TAK-831 500 mg vs Part 1: TAK-831 750 mg; Dose proportionality was evaluated using the following power model: ln (PK Parameter) is equal to (=) a+b*ln (dose), where a and b are the intercept and slope of the line, respectively. Dose proportionality was declared when the 90 percent (%) confidence interval (CI) of the slope lies entirely within the critical region (0.9483, 1.0517) for the dose range of 10 mg to 750 mg; Test type: Superiority or Other; Slope = 0.6662, 90% CI 2-sided [0.5969 to 0.7355]
Statistical Analysis 2: Comparison: Part 2: TAK-831 30 mg vs Part 2: TAK-831 100 mg vs Part 2: TAK-831 200 mg vs Part 2: TAK-831 400 mg; Dose proportionality was evaluated using the following power model: ln (PK Parameter) = a+b*ln (dose), where a and b were the intercept and slope of the line, respectively. Dose proportionality was declared when the 90% CI of the slope lies entirely within the critical region (0.9139, 1.0861) for the dose range of 30 mg to 400 mg; Test type: Superiority or Other; Power model; Slope = 0.7795, 90% CI 2-sided [0.6597 to 0.8993]
Statistical Analysis 3: Comparison: Part 4: TAK-831 100 mg Tablet Fasted vs Part 4: TAK-831 100 mg Suspension Fasted; The point estimate and CI were obtained by taking the antilog of the difference in the log transformed lease square (LS) Means; Test type: Superiority or Other; Least Square (LS) Mean Ratio = 0.362, 90% CI 2-sided [0.3043 to 0.4301]
Statistical Analysis 4: Comparison: Part 4: TAK-831 100 mg Tablet Fasted vs Part 4: TAK-831 100 mg Tablet Fed; The point estimate and CI were obtained by taking the antilog of the difference in the log transformed LS Means; Test type: Superiority or Other; LS Mean Ratio = 1.799, 90% CI 2-sided [1.4625 to 2.2116]

6. Secondary Outcome: Part 2 and 3: Cmax, ss: Maximum Observed Plasma Concentration at Steady State for TAK-831
Time Frame: Day 16 (Part 2) and Day 14 (Part 3) pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK set included all participants with at least 1 estimable PK parameter for TAK-831. Due to discomfort observed in participants from the CSF collection procedure, Part 3 of the study was terminated hence no participants were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: TAK-831 400 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
ng/mL | 177.5 (45.85) | 560.7 (214.90) | 897.7 (192.73) | 1269.5 (451.37) |

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours in Part 1 and up to 72 hours in Part 2 and 4) post-dose; Day 16 (Part 2) and Day 14 (Part 3) pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 23 | 23 | 24
hours
  Day 1 | 0.250 [0.23 to 0.50] | 0.260 [0.25 to 0.33] | 0.435 [0.23 to 1.50] | 0.275 [0.23 to 2.02] | 0.725 [0.20 to 1.00] | 0.760 [0.25 to 2.02] | 0.500 [0.47 to 0.68] | 0.500 [0.17 to 2.00] | 0.375 [0.17 to 1.02] | 0.500 [0.15 to 1.00] |  |  | 0.930 [0.25 to 4.00] | 3.980 [0.95 to 4.05] | 0.250 [0.17 to 2.02]
  Day 16 | NA [NA to NA] — Tmax for Part 1 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 1 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 1 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 1 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 1 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 1 was not planned to analyzed on Day 16. | 0.500 [0.48 to 0.53] | 0.365 [0.23 to 0.98] | 0.500 [0.20 to 0.50] | 0.490 [0.23 to 1.00] |  |  | NA [NA to NA] — Tmax for Part 4 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 4 was not planned to analyzed on Day 16. | NA [NA to NA] — Tmax for Part 4 was not planned to analyzed on Day 16.

8. Secondary Outcome: Part 1, 2 and 4: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours in Part 1 and up to 72 hours in Part 2 and 4) post-dose
Population: The PK set included all participants with at least 1 estimable PK parameter for TAK-831.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 23 | 23 | 24
nanogram*hour per milliliter (ng*hr/mL) | 98.0 (17.02) | 463.8 (80.13) | 1186.8 (256.67) | 1900.8 (293.72) | 4111.1 (1599.18) | 5374.0 (1651.36) | 296.3 (95.31) | 938.4 (180.29) | 2030.2 (265.73) | 2832.7 (819.36) | 598.6 (310.31) | 1397.7 (434.45) | 1083.6 (302.13)
Statistical Analysis 1: Comparison: Part 1: TAK-831 10 mg vs Part 1: TAK-831 30 mg vs Part 1: TAK-831 100 mg vs Part 1: TAK-831 250 mg vs Part 1: TAK-831 500 mg vs Part 1: TAK-831 750 mg; Dose proportionality was evaluated using the following power model: ln (PK Parameter) = a+b*ln (dose), where a and b are the intercept and slope of the line, respectively. Dose proportionality was declared when the 90 % CI of the slope lies entirely within the critical region (0.9483, 1.0517) for the dose range of 10 mg to 750 mg; Test type: Superiority or Other; Slope = 0.8720, 90% CI 2-sided [0.8145 to 0.9296]
Statistical Analysis 2: Comparison: Part 2: TAK-831 30 mg vs Part 2: TAK-831 100 mg vs Part 2: TAK-831 200 mg vs Part 2: TAK-831 400 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; Power model; Slope = 0.9135, 90% CI 2-sided [0.8062 to 1.0209]
Statistical Analysis 3: Comparison: Part 4: TAK-831 100 mg Tablet Fasted vs Part 4: TAK-831 100 mg Suspension Fasted; The point estimate and CI were obtained by taking the antilog of the difference in the log transformed LS Means; Test type: Superiority or Other; LS Mean Ratio = 0.500, 90% CI 2-sided [0.4324 to 0.5777]
Statistical Analysis 4: Comparison: Part 4: TAK-831 100 mg Tablet Fasted vs Part 4: TAK-831 100 mg Tablet Fed; The point estimate and CI were obtained by taking the antilog of the difference in the log transformed LS Means; Test type: Superiority or Other; LS Mean Ratio = 2.563, 90% CI 2-sided [2.1000 to 3.1275]

9. Secondary Outcome: Part 1, 2 and 4: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours in Part 1 and up to 72 hours in Part 2 and 4) post-dose
Population: The PK set included all participants with at least 1 estimable PK parameter for TAK-831.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 23 | 23 | 24
ng*hr/mL | 109.7 (22.02) | 499.2 (92.57) | 1271.4 (253.26) | 1945.5 (294.36) | 4140.7 (1602.32) | 5512.0 (1721.84) | 342.9 (46.80) | 980.5 (204.04) | 2092.7 (273.06) | 2866.6 (822.22) | 653.7 (308.86) | 1428.8 (433.24) | 1115.3 (296.56)
Statistical Analysis 1: Comparison: Part 1: TAK-831 10 mg vs Part 1: TAK-831 30 mg vs Part 1: TAK-831 100 mg vs Part 1: TAK-831 250 mg vs Part 1: TAK-831 500 mg vs Part 1: TAK-831 750 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, Power model; Slope = 0.8505, 90% CI 2-sided [0.7925 to 0.9084]
Statistical Analysis 2: Comparison: Part 2: TAK-831 30 mg vs Part 2: TAK-831 100 mg vs Part 2: TAK-831 200 mg vs Part 2: TAK-831 400 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, Power model; Slope = 0.8415, 90% CI 2-sided [0.7618 to 0.9212]
Statistical Analysis 3: Comparison: Part 4: TAK-831 100 mg Tablet Fasted vs Part 4: TAK-831 100 mg Suspension Fasted; The point estimate and CI were obtained by taking the antilog of the difference in the log transformed LS Means; Test type: Superiority or Other; LS Mean Ratio = 0.543, 90% CI 2-sided [0.4797 to 0.6149]
Statistical Analysis 4: Comparison: Part 4: TAK-831 100 mg Tablet Fasted vs Part 4: TAK-831 100 mg Tablet Fed; The point estimate and CI were obtained by taking the antilog of the difference in the log transformed LS Means; Test type: Superiority or Other; LS Mean Ratio = 2.336, 90% CI 2-sided [1.9592 to 2.7854]

10. Secondary Outcome: Part 2 and 3: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-831
Time Frame: Day 16 (Part 2) and Day 14 (Part 3) pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: TAK-831 400 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
ng*hr/mL | 319.8 (83.06) | 1211.0 (236.45) | 1973.0 (316.34) | 3452.6 (1249.58) |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Part 1 Day 31, Part 2 Day 46, Part 3 Day 44 and Part 4 Day 43)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Placebo Pooled | Part 1: TAK-831 10 mg | Part 1: TAK-831 30 mg | Part 1: TAK-831 100 mg | Part 1: TAK-831 250 mg | Part 1: TAK-831 500 mg | Part 1: TAK-831 750 mg | Part 2: Placebo Pooled | Part 2: TAK-831 30 mg | Part 2: TAK-831 100 mg | Part 2: TAK-831 200 mg | Part 2: TAK-831 400 mg | Part 3: Placebo | Part 3: TAK-831 400 mg | Part 4: TAK-831 100 mg Tablet Fasted | Part 4: TAK-831 100 mg Tablet Fed | Part 4: TAK-831 100 mg Suspension Fasted
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/1 | 0/5 | 0/23 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 6/12 | 2/6 | 2/6 | 2/6 | 1/6 | 3/6 | 4/6 | 6/8 | 5/6 | 6/6 | 2/6 | 5/6 | 1/1 | 5/5 | 5/23 | 3/23 | 4/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo Pooled (N=12) | Part 1: TAK-831 10 mg (N=6) | Part 1: TAK-831 30 mg (N=6) | Part 1: TAK-831 100 mg (N=6) | Part 1: TAK-831 250 mg (N=6) | Part 1: TAK-831 500 mg (N=6) | Part 1: TAK-831 750 mg (N=6) | Part 2: Placebo Pooled (N=8) | Part 2: TAK-831 30 mg (N=6) | Part 2: TAK-831 100 mg (N=6) | Part 2: TAK-831 200 mg (N=6) | Part 2: TAK-831 400 mg (N=6) | Part 3: Placebo (N=1) | Part 3: TAK-831 400 mg (N=5) | Part 4: TAK-831 100 mg Tablet Fasted (N=23) | Part 4: TAK-831 100 mg Tablet Fed (N=23) | Part 4: TAK-831 100 mg Suspension Fasted (N=24)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (3) | 4 (7) | 0 (0) | 2 (3) | 1 (2) | 5 (16) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 3 (7) | 4 (13) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.